CLINICAL TRIAL: NCT05266482
Title: Personal Feedback on Patient-reported Outcomes to Fulfil or Exceed Preoperative Expectations of Primary Total Knee Arthroplasty Patients: PAK-study.
Brief Title: Personalized Information Before and After Total Knee Arthroplasty: PAK-study
Acronym: PAK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kliniek ViaSana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N21.077
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Total Knee Arthroplasty
Keywords: Satisfaction; Expectations; Personal feedback
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Next to the usual care, patients also get the opportunity to download and read a personal report.
  Interventions: Other: Personal report
- Control group (No Intervention): Patients will receive the usual care.

INTERVENTIONS:
Other: Personal report — In the intervention group, in addition to receiving the usual care, patients will receive personal reports on multiple time points. These reports include feedback on their PROs including reference scores of patients who previously underwent total knee replacement surgery.
  Arms: Intervention group

SUMMARY:
Despite positive results following total knee arthroplasty (TKA), some patients are dissatisfied after recovery. Unfulfilled expectations is a key predictor of dissatisfaction. The aim of this study is to investigate if more patients fulfil or exceed their preoperative expectations one year after TKA when personal feedback on their PROs is given.

ELIGIBILITY:
Inclusion Criteria:

* Planned for primary TKA in Kliniek ViaSana
* Signed informed consent

Exclusion Criteria:

* Aged under 18 years
* Do not possess an own email adress,
* Do not have a thorough command of the Dutch language,
* Previously received contra-lateral primary TKA and/or unicompartmental KA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Patients' expectations | 12 months after surgery
  The percentage (0%-100%) of patients who fulfil or exceed their preoperatively set expectations 12 months after TKA surgery. Measured using HSS-KRES.

SECONDARY OUTCOMES:
Patients' expectations | 3 and 6 months after surgery
  The percentage (0%-100%) of patients who fulfil or exceed their preoperatively set expectations 3 and 6 months after TKA surgery. Measured using HSS-KRES.
Patients' satisfaction | 3, 6 and 12 months after surgery
  Satisfaction score with the outcome of TKA surgery. Measured using NRS satisfaction from 0 (dissatisfied) to 10 (satisfied).
Pain relief | 3, 6 and 12 months after surgery
  Measured on a scale from 1 (very much deteriorated) to 7 (very much improved)
Functional improvement | 3, 6 and 12 months after surgery
  Measured on a scale from 1 (very much deteriorated) to 7 (very much improved)
Perceived recovery | 3, 6 and 12 months after surgery
  Measured on a scale from 0 (worse than ever) to 6 (fully recovered)

CONTACTS AND LOCATIONS:
Overall Officials: J.M. Brinkman, MD, PhD, Principal Investigator — Kliniek ViaSana
Locations (1):
- Kliniek ViaSana, Mill, Netherlands

IPD SHARING:
Plan to Share IPD: No